CLINICAL TRIAL: NCT05359406
Title: Radiotherapy Followed by Chemotherapy With Target Therapy and Anti-PD-1 Immunotherapy in Locally Advanced Rectal Cancer With Refractory Liver Metastasis/Pulmonary Metastasis(Miracle-2): A Prospective, Single Arm, Multi-Center, Phase II Clinical Trial
Brief Title: A Combination Therapy Including Anti-PD-1 Immunotherapy in Rectal Cancer With Refractory Distal Metastasis
Acronym: Miracle-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LI XIN-XIANG (Other)
Responsible Party: Sponsor-Investigator, LI XIN-XIANG, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Miracle-2
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Advanced Rectal Cancer; Distal Metastasis
Keywords: anti-PD-1 immunotherapy; short-course radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unresectable group (Experimental): Patients will receive tislelizumab in combination with radiotherapy and targeted therapy. 2 weeks after large fractionated radiotherapy for primary rectum lesion and metastasis, patients will be treated with systemic treatment including chemotherapy combined with targeted therapy and immunotherapy. Patients will be evaluated by MDT every 2 months since the beginning of the treatment. Those who are regarded as NED will be treated surgically/locally. Those in stable or partial remission will continue with combination therapy. Those with progressive disease will be withdrawn from study. Patients who are not surgically treatable will continue with combination therapy until disease progression or receiving surgical treatment.
  Interventions: Combination Product: a combination therapy including tislelizumab

INTERVENTIONS:
Combination Product: a combination therapy including tislelizumab — For liver/pulmonary metastasis, the treatment plan is to implement large fraction radiotherapy for 4-8 times. For primary rectum lesion, short-course radiotherapy regimen through intensity-modulated radiotherapy will be applied with dose of 25Gy/5Fx. Immunotherapy contains anti-PD-1 monoclonal antibody, Tislelizumab(200mg, d1, q3w, i.v). For patients with RAS or BRAF mutation, chemotherapy adopts FOLFOX+BEV plan. For patients without RAS or BRAF mutation, chemotherapy adopts FOLFIRI+CET plan.
  Patients will be followed for safety during the study. The safety follow-up period is defined as 90 days after the last dose of tislelizumab. Safety related data will be collected from the time of signing the informed consent until the end of the safety follow-up period or the start of new therapy.
  Other Names: Radiotherapy Followed by Chemotherapy with target therapy and anti-PD-1 immunotherapy

SUMMARY:
Though surgical resection remains the primary choice for advanced rectal cancer, about 80% are considered unresectable due to the number, size, or location of metastases. The overall prognosis of patients who accepted traditional treatment methods is still poor. Therefore, the investigators designed a combination therapy, short-course radiotherapy followed by chemotherapy with target therapy and anti-PD-1 immunotherapy. This study implement the combination therapy in patients with rectal cancer who are initially unresectable in the locally advanced stage with multiple liver/pulmonary metastases, to evaluate whether they can improve the objective response rate, the conversion rate of radical surgery and prolong the overall survival of patients, and strive to provide high-level medical evidence for the clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~70;
* Patient signs informed consent;
* ECOG score 0~1;
* Initial colonoscopy and pathology: adenocarcinoma;
* MRI: rectal cancer located less than 10cm from the anus;
* Imaging confirms multiple measurable metastases exist in the liver or lung , which are evaluated as NED unacceptable by MDT discussion;
* no previous treatment;
* Patients have adequate organ function;
* No contraindications to surgery or chemoradiation;
* The relevant test results within 7 days before the first dose must meet the following requirements:

  1. Blood routine examination (no blood transfusion within 7 days before screening, no correction with hematopoietic stimulating factor drugs):

     * Hb≥90g/L
     * ANC≥1.5×10^9/L; LC≥0.5×10^9/L;
     * PLT≥100×10^9/L;
     * WBC≥3.0×10^9/L, ≤15×10^9/L;
  2. Blood chemistry (no blood transfusion or albumin within 7 days prior to screening):

     * ALT, AST≤1.5 ULN;
     * ALP≤2.5 ULN;
     * TBIL≤1.5 ULN;
     * Cr≤1.5 ULN, CrCL≥50 mL/min;
     * PT, APTT≤1.5 ULN, INR≤1.5 ULN(not receiving anticoagulation);
  3. TSH is within the normal range; if TSH is out of the normal range, FT3 and FT4 should be investigated. If the test results of FT3/FT4 cannot be obtained, T3 and T4 can be accepted. If the level of T3/T4 is normal, the patients can be selected.
  4. Urine test: urine protein<2+; if the urine protein≥2+, the 24-hour urine protein quantification must be≤1g;
  5. Echocardiography: LVEF≥55%;
  6. 12-lead ECG: Fridericia corrected QTcF<470 msec.
* Expected survival time >6 months;
* The gene status of KRAS, NRAS, BRAF and HER2 is clear;
* Patients are willing and able to follow the protocol during the study, including receiving treatment and scheduled follow-up and examination.

Exclusion Criteria:

Patients will not be accepted into this study if they meet any of the following criteria:

1. History of tumor-related disease and treatment:

1. Age <18 or >75 years;
2. other malignancy within 5 years, except adequately treated carcinoma in situ of the cervix or squamous cell carcinoma of the skin, or largely controlled basal cell carcinoma of the skin;
3. malignant pleural effusion or malignant ascites;
4. patients with severe medical comorbidities that preclude radiotherapy and surgery;
5. previously treated;
6. clinical or radiological evidence of spinal cord compression or a tumor within 3mm of the spinal cord on MRI
7. the presence of distant metastases besides the liver and lungs, including brain, bone, ovarian, peritoneal and retroperitoneal multiple lymph node metastases;
8. Patients who are considered suitable for using intense systemic treatment to achieve conversion after MDT discussion;
9. pathological diagnosis of indolent cell carcinoma;
10. patients with microsatellite instability or dMMR;
11. patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. that require emergency surgical resection;

2. Co-morbidities and treatment history:

1. Presence of immunodeficiency disorders, including primary immunodeficiency disorders (e.g. caused by genetic factors) or secondary immunodeficiency disorders (e.g. caused by HIV infection or treatment related to immunological agents, etc.);
2. Presence of any autoimmune disease that still requires treatment or a previous history of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, rheumatic heart valve disease, glomerulonephritis, etc. Excluding hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement therapy and type I diabetes with manageable and stable blood glucose;
3. known or suspected interstitial pneumonia; other moderate to severe lung disease that may interfere with the detection or management of drug-related pulmonary toxicity and severely affect respiratory function, including idiopathic pulmonary tissue fibrosis, mechanized pneumonia/occlusive fine bronchitis, etc.;
4. severe cardiovascular disease, including but not limited to conditions meeting NYHA criteria (Class III or higher), or myocardial infarction or cerebrovascular accident (cerebral ischaemia, symptomatic cerebral infarction, etc.) occurring within 3 months prior to the first dose, or unstable arrhythmia or unstable angina pectoris with coronary artery disease occurring within 1 month prior to the first dose, or congestive heart failure, or pre-existing symptomatic superior vena cava syndrome, etc.;
5. an arteriovenous thrombotic event, such as deep vein thrombosis and pulmonary embolism, within the previous 3 months;
6. history of live attenuated vaccination within 28 days prior to the first study dose or anticipated need for live attenuated vaccination during the study;
7. active hepatitis B (defined as positive hepatitis B virus surface antigen [HBsAg] test result and HBV-DNA test value ≥ 500 IU/ml);
8. Hepatitis C (defined as a positive test result for hepatitis C virus antibody [HCV-Ab]) ;
9. history of tuberculosis infection or treatment within 1 year prior to signing informed consent;
10. presence of severe infection within 4 weeks prior to first dose, including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc.; or active infection requiring systemic antibiotic therapy according to NCI-CTCAE v5.0 grade ≥ 2 within 2 weeks prior to first dose, or unexplained fever >38.5°C during screening/prior to first dose (at the investigator's discretion, due to oncologic causes fever due to tumor causes may be enrolled);
11. previous allogeneic bone marrow transplantation or solid organ transplantation received or intended to be received;
12. Hemoptysis with a maximum daily hemoptysis of approximately ≥2.5 ml within 2 months prior to signing informed consent; clinically significant bleeding symptoms or a clear bleeding tendency within 1 month prior to signing informed consent, e.g. gastrointestinal bleeding, bleeding gastric ulcer, fecal occult blood ++ at baseline, vasculitis; known hereditary or acquired bleeding and thrombotic tendencies, e.g. hemophilia, impaired coagulation skills, thrombocytopenia, hypersplenism, etc.;
13. abnormal coagulation (INR > 1.5 or APTT > 1.5 × ULN) with bleeding tendency or undergoing thrombolysis or requiring long-term anticoagulation with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day)
14. peripheral neuropathy ≥ grade 2 according to NCI-CTCAE v5.0;
15. Co-morbidities of other infectious diseases that are not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Early Tumor Shrinkage | 5 years after intervention
  The relative change of the sum of the longest diameters of the baseline RECIST target lesion at 8 weeks of systemic therapy, distinguished by 20% as the cut-off point between early response and no response.

SECONDARY OUTCOMES:
Disease Control Rate | 5 years after intervention
  Percentage of patients with disease control in non-irradiated metastatic lesions
Duration of Response | 5 years after intervention
  The time between PR/CR and subsequent progressive disease or death of any cause.
Overall Survival | 5 years after intervention
  The time from the beginning of treatment to the date of death.
Progression-Free Survival | 5 years after intervention
  The time from the start of treatment to PD or death of any cause.
Acute toxicity associated with immunotherapy | from the beginning of the treatment to 90 days after the end of immunotherapy
  Proportion of patients with treatment-related acute toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinxiang Li, Shanghai, Shanghai Municipality, China